CLINICAL TRIAL: NCT06817577
Title: A First-in-human (FIH) Clinical Trial to Investigate the Human Monoclonal Antibody NG004, Administrated Intrathecally in Acute Spinal Cord Injury (SCI) Patients
Brief Title: NG004 in Spinal Cord Injury Patients
Acronym: SPROUT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NovaGo Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NG004-SCI-001; 2024-514303-34-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-13; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Acute Spinal Cord Injury (SCI); Spinal Cord Diseases; Central Nervous System Diseases; Nervous System Diseases; Trauma, Nervous System; Spinal Cord Injuries (SCI); Wounds and Injuries
Keywords: Acute spinal cord injury; Nogo-A; SPROUT; Regeneration
MeSH Terms: conditions — Spinal Cord Diseases; Central Nervous System Diseases; Nervous System Diseases; Trauma, Nervous System; Spinal Cord Injuries; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NG004 (Experimental)
  Interventions: Drug: NG004

INTERVENTIONS:
Drug: NG004 — repeated intrathecal injections of NG004

SUMMARY:
This is the FIH, multicenter, open-label, sequential, multiple ascending dose trial of NG004 in patients with acute incomplete cervical SCI. The trial will evaluate the safety, tolerability, and PK of 4 dose regimens of NG004, and will evaluate the maximum tolerated dose of NG004.

ELIGIBILITY:
Inclusion Criteria:

* Acute incomplete cervical SCI (Neurological level of injury C1 ≤ lesion ≤ C8) with confirmed classification of American Spinal Injury Association (ASIA) impairment scale (AIS) C-D at Screening
* 4-28 days post-injury
* No required mechanical ventilation or patients that not completely depend on mechanical ventilation
* Hemodynamically and clinical stable patient according to the acute SCI condition at baseline

Exclusion Criteria:

* Trauma caused by ballistic or other injury that directly penetrates the spinal cord including gunshot and knife wounds
* Multiple levels of clinically relevant spinal cord lesions
* Major brachial or lumbar plexus damage/trauma
* Significant head trauma or other injury that was, in the opinion of the investigator, sufficient to interfere with the assessment of the spinal cord function
* Other significant pre-existing or current severe systemic disease such as lung, liver (exception: history of uncomplicated Hepatitis A), gastrointestinal, cardiac, immunodeficiency (including anamnestic known HIV) or kidney disease; or active malignancy
* History of or an acute episode of Multiple Sclerosis or Guillain-Barre syndrome History of recent (6 months) meningitis or meningoencephalitis
* History of refractory epilepsy
* History of or current autoimmune disease
* Patients with uncontrolled bleeding diathesis and/or who require concomitant therapeutic anticoagulation and not related to SCI
* Presence of any unstable medical or psychiatric condition
* Drug dependence any time during the 6 month's preceding trial entry
* Pregnant or nursing women
* History of a life-threatening allergic or immune mediated reaction
* Patients with the presence of infection around the location where the spinal needle insertions are planned for applying the intrathecal injections
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations
* Patients who are unconscious

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Type, frequency, severity, and causal relationship of adverse events (AEs), serious AEs, and adverse drug reactions | From treatment start up to 6 months

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] in serum | After first and last intrathecal injection, measured at pre-dose and 1, 3, 6, 24, 48 hours post-dose.
Half-life in serum [T1/2] | After last intrathecal injection up to 6 months

OTHER OUTCOMES:
Effect on motor function as Change from Baseline in ISNCSCI upper extremities motor score (UEMS), according to the International Standards for the Neurological Classification of Spinal Cord Injury (ISNCSCI) protocol | Baseline up to 6 months
  The ISNCSCI bilateral Upper Extremity Motor Score (UEMS) is determined by examining the muscle function within each of the 5 myotomes encompassing arm and hand function on each side of the body. A score ranging from 0 to 5 can be given to each myotome tested resulting in a maximum score of 50. Higher values indicate better recovery.
Effect on daily life functioning according to change in Version III of the Spinal Cord Independence Measure (SCIM-III) | Baseline to 6 months
  The SCIM III questionnaire self-care score assesses activities of daily living including feeding, bathing, dressing, and grooming. The self-care score ranges 0-20. The higher scores correspond to better ability to carry out the self-care activities.

CONTACTS AND LOCATIONS:
Overall Officials: Director of Clinical Research, Study Director — NovaGo Therapeutics AG
Locations (6):
- Germany (4):
  - Klinik für Querschnittgelähmte, Klinikum Bayreuth, Bayreuth
  - Zentrum für Rückenmarkverletzte und Klinik für Orthopädie, BG Klinikum Bergmannstrost, Halle
  - Klinik für Paraplegiologie, Universitätsklinikum Heidelberg, Heidelberg
  - Zentrum für Rückenmarksverletzte, Unfallklinik Murnau, Murnau am Staffelsee
- Switzerland (2):
  - Swiss Paraplegic Centre, Nottwil
  - Universitätsklinik Balgrist, Zurich

IPD SHARING:
Plan to Share IPD: No